CLINICAL TRIAL: NCT03023501
Title: The Effect of Gabapentin on Postoperataive Pain ,Morphine Sparing Effect and Preoperative Anxiety in Bariatric Surgical Patients
Brief Title: Effect of Gabapentin on Postoperative Morphine Consumption After Sleeve Gastrectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, MUEEN ULLAH KHAN, MUEEN ULLAH KHAN, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-13-902
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin (Experimental): Gabapentin 1200mg capsule was administered orally 2 hours before surgery
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Placebo capsule was prepared by hospital pharmacy and was administered orally 2 hours before surgery.
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Gabapentin
  Arms: Gabapentin
Drug: Placebo Oral Capsule
  Arms: Placebo

SUMMARY:
The evidence regarding effects of pain modulator like gabapentin on postoperative pain after sleeve gastrctomy is sparse. Gabapentin has anti-hyperalgesic and postoperative opioid-sparing properties.This study will highlight the effectiveness of preoperative use of gabapentin for postoperative pain management in morbidly obese patients.

DETAILED DESCRIPTION:
Research Problem: Laprocopic sleeve gastrectomy is the most common surgical procedure performed for reducing weight in morbidly obese patients. Laparoscopic surgery is considered to be less invasive than open surgery. The treatment of pain in obese patients is a challenge. Administering opioids, can have an increasing effect of respiratory depression in patients already at risk of sleep apnea. The evidence regarding effects of pain modulator like gabapentin on postoperative pain after sleeve gastrctomy is sparse. Gabapentin has anti-hyperalgesic and postoperative opioid-sparing properties. The analgesic effect of gabapentin appears to be related to the surgical procedure undertaken, a more procedure-specific evaluation is needed for different types of surgeries..

Research Significance: This study will highlight the effectiveness of preoperative use of gabapentin for postoperative pain management in morbidly obese patients.

Research Objectives: To evaluate the effect of preoperative administration of gabapentin on postoperative pain, postoperative morphine consumption and preoperative anxiety in patients coming for laparoscopic sleeve gastrectomy.

Research Methodology:

Inclusion criteria: ASA I and II, Age 18-50 years, either sex, Planned Surgical procedure laparoscopic sleeve garstectomy, BMI 30-45 . Exclusion criteria: Patients taking any sedative, tranquillizers , history of sleep apnoea ,contraindications to gabapentin, Methods Patients will be randomly assigned into two groups, Group-Control and , Group- Gabapentin of 25 each. Anesthesia and postoperative course will be standardized. VAS scale will be used for assessment of preoperative anxiety and postoperative pain. Post operatively pain assessment and morphine consumption will be performed for 24 hours in PACU and ward

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and 2
* BMI 35 - 45

Exclusion Criteria:

* Patients taking any sedative or tranquillizers
* Any contraindication to gabapentin.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Post operative Morphine requirement | At 2 hours in Post Anesthesia Care Unit
Post operative pain | At 2 hours in Post Anesthesia Care Unit
Post operative Morphine requirement | 4 hourly in the ward for 24 hours
Post operative pain | 4 hourly in the ward for 24 hours

SECONDARY OUTCOMES:
Preoperative anxiety | 30 minutes before surgery

IPD SHARING:
Plan to Share IPD: Yes